CLINICAL TRIAL: NCT04774211
Title: Prospective Prevalence and Validation Study of Pediatric Intensive Care Delirium.
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Rikke Louise Stenkjær, Principal investigator, Rigshospitalet, Denmark
Other Study IDs: NNF20OC0066074
Record Dates: First submitted 2021-02-22; First posted 2021-03-01 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Pediatric Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: SOS-PD — Validation of SOS-PD bedside assessments comparing the Danish SOS-PD scale with a Child Psychiatrist using DSM-V as the reference standard

SUMMARY:
Pediatric delirium (PD) is a poorly investigated clinical problem that needs to be further explored in a Danish context. Children are at risk of discomfort and suffering if they experience delirium. The condition is associated with prolonged mechanical ventilation, longer hospital stay, increased mortality, and risk of long-term cognitive impairment. Therefore, it is important to assess critically ill children with a validated tool to enable early detection and management of the condition. In this study, the investigators will determine the prevalence of pediatric intensive care delirium. To this end, the investigators will validate the Sophia Observation withdrawal Symptoms - Pediatric delirium scale (SOS-PD) for patient assessment.

DETAILED DESCRIPTION:
Prospective prevalence and validation study of pediatric intensive care delirium.

Aim: To validate the SOS-PD assessment tool and determine the prevalence of delirium in children aged 3 months to 18 years in a Danish context.

Data analysis and power calculation: With 140 patients, the accuracy estimate in this study will have a 95% confidence interval of +/- 5%. Accuracy defined as (true positive + true negative) / all x 100 is expected to be 90%. The validity of the SOS-PD assessment tool is calculated from standard definitions of sensitivity, specificity, positive predictive value and negative predictive value. The prevalence is calculated in percent. All data will be entered and encoded in RedCap and exported to SPSS for statistical analysis of data.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric intensive care patients
* Length of stay of 48 hours or more

Exclusion Criteria:

* Non Danish speaking
* Use of neuromuscular blocking agents
* sedation level at COMFORT behavior score > 11 or Richmond Agitation Sedation Scale > -3

Ages: 3 Months to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Pediatric intensive care patients
Sampling Method: Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of delirium in children aged 3 months -18 years of age | The observation period is 24 hours
  Delirium prevalence is determined by the proportion of patients that had at least one positive delirium score with patients that never had a positive delirium score determined by Sophia Observation Withdrawal Symptoms - Pediatric Delirium scale (SOS-PD). The minimum score of SOS-PD is 0 and maximum score is 17. The score ≥4 indicates delirium.

SECONDARY OUTCOMES:
Validation of the Sophia Observation Withdrawal Symptoms - Pediatric Delirium scale (SOS-PD) assessment tool in to a Danish context. | The observation period is 24 hours
  The validity of the SOS-PD assessment tool is calculated from standard definitions of sensitivity, specificity, positive predictive value and negative predictive value

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Forsyth Herling, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No